CLINICAL TRIAL: NCT00356941
Title: Phase I Study of Oxaliplatin in Combination With Docetaxel and Radiotherapy in Patients With Unresectable or Recurrent Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Oxaliplatin, Docetaxel, and Radiation Therapy in Treating Patients With Unresectable Stage II/III or Recurrent NSCLC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Withdrawn due to lack of accrual
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Chinsoo Cho MD, Masonic Cancer Center, University of Minnesota
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005LS073; UMN-0511M77529 (Other: IRB, University of Minnesota); UMN-OX-04-007 (Other: Sanofi Research Division)
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Oxaliplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemoradiation Treated Patients (Experimental): Patients receiving Docetaxel, Oxaliplatin and radiotherapy.
  Interventions: Drug: docetaxel; Drug: oxaliplatin; Procedure: radiation therapy

INTERVENTIONS:
Drug: docetaxel — 60 mg/m2 on day 1 of each week during radiation therapy
  Other Names: Taxotere
Drug: oxaliplatin — Escalating dose per assignment: 20-50 mg/m2 on day 2 of each week during radiation therapy
  Other Names: Eloxatin
Procedure: radiation therapy — 2 Gy Days 1-5 each week, total dose of 70Gy
  Other Names: radiotherapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as oxaliplatin and docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Oxaliplatin and docetaxel may make tumor cells more sensitive to radiation therapy. Giving oxaliplatin and docetaxel together with radiation therapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of oxaliplatin when given together with docetaxel and radiation therapy in treating patients with unresectable stage II or stage III or recurrent non-small cell lung cancer .

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of oxaliplatin when given with docetaxel and thoracic radiotherapy in patients with unresectable stage II, IIIA, or IIIB or recurrent non-small cell lung cancer.

Secondary

* Determine the dose-limiting toxicities of this regimen in these patients.
* Determine the objective tumor response in patients treated with this regimen.

OUTLINE: This is a dose-escalation study of oxaliplatin.

* Induction therapy: Patients undergo radiotherapy once a day on days 1-5, 8-12, 15-19, 22-26, 29-33, 36-40, and 43-47. Patients also receive docetaxel intravenous (IV) over 1 hour on days 1, 8, 15, 22, 29, 36, and 43 and oxaliplatin IV over 2-4 hours on days 2, 9, 16, 23, 30, 37, and 44. Patients with stable or responding disease proceed to consolidation therapy.

Cohorts of 6 patients receive escalating doses of oxaliplatin during induction therapy until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 3 of 6 patients experience dose-limiting toxicity.

* Consolidation therapy: Beginning 3 weeks after the completion of induction therapy, patients receive consolidation therapy comprising docetaxel IV over 1 hour immediately followed by oxaliplatin IV over 2-4 hours on day 1. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 4 weeks and then every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-small cell lung cancer (NSCLC) meeting 1 of the following criteria:

  * Medically inoperable or unresectable stage II, IIIA, or IIIB disease
  * Post-resection intrathoracic tumor recurrence
* Measurable disease by computed tomography(CT) scan
* No evidence of small cell histology
* No significant pleural effusion on chest x-ray or malignant pleural effusion on cytology
* No metastatic disease
* Eastern Cooperative Oncology Group (ECOG) (Zubrod) performance status 0-1
* Absolute granulocyte count ≥ 2,000/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 8.0 g/dL
* Bilirubin ≤ 1.5 mg/dL
* Serum glutamic oxaloacetic transaminase (SGOT) ≤ 1.5 times upper limit of normal (unless abnormality is caused by documented benign disease)
* Creatinine ≤ 1.5 mg/dL
* Weight loss ≤ 10% within the past 3 months
* Forced expiratory volume (FEV) 1 ≥ 1,000 cc
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment

Exclusion Criteria:

* Synchronous (except for nonmelanomatous skin cancer) or prior invasive malignancy, unless disease free for > 3 years
* Myocardial infarction within the past 6 months
* Symptomatic heart disease, including any of the following:

  * Angina
  * Congestive heart failure
  * Uncontrolled arrhythmia
* Active infection or fever ≥ 38.5°C within the past 3 days
* Known hypersensitivity to any of the components of oxaliplatin or docetaxel
* Prior thoracic or neck radiotherapy
* Prior docetaxel or oxaliplatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-04; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of oxaliplatin in combination with docetaxel and radiotherapy | Within 90 days of radiotherapy

SECONDARY OUTCOMES:
Dose-limiting toxicities | Within 90 days of radiotherapy
Objective tumor response | Every 3 months up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: L. Chinsoo Cho, MD, Study Chair — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of Minnesota Cancer Center, Minneapolis, Minnesota, United States